CLINICAL TRIAL: NCT05276674
Title: Post-Market Clinical Follow-up Study on the ZNN™ Bactiguard ® Retrograde Femoral Nails (Implants and Instrumentation)
Brief Title: ZNN Bactiguard Retrograde Femoral Nails PMCF Study
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2021-40T
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Femoral Fracture
Keywords: Bactiguard; Femur fracture; Intramedullary nailing; Infection control
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ZNN Bactiguard Retrograde Femoral Nail: Patients implanted with a ZNN Bactiguard Retrograde Femoral Nail for fixing and stabilizing a femoral fracture.
  Interventions: Device: ZNN Bactiguard Retrograde Femoral Nail

INTERVENTIONS:
Device: ZNN Bactiguard Retrograde Femoral Nail — Femoral fracture internal fixation.

SUMMARY:
Post-market clinical follow-up (PMCF) study to confirm the safety, performance, and clinical benefits of the intra-medullary retrograde femoral nail Zimmer Natural Nail (ZNN) Bactiguard (implants and instrumentation) when used for the temporary internal fixation and stabilization of femoral fractures.

DETAILED DESCRIPTION:
The objective of this prospective PMCF study is to collect data to confirm safety, performance and clinical benefits of the Zimmer Natural Nail (ZNN) Bactiguard Retrograde Femoral Nail (implants and instrumentation) when used for the temporary internal fixation and stabilization of femoral fractures.

The primary endpoint is the assessment of performance by analyzing fracture healing.

The secondary endpoints are the assessment of safety, clinical benefit and post-op fracture related infection (FRI). Safety will be evaluated by recording and analyzing the incidence and frequency of complications and adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified. Clinical benefit will be assessed by recording patient-reported outcome measures (PROMs). FRIs will be classified according to the updated diagnostic algorithm defined by the FRI Consensus Group.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older.
* Patient must have a femoral fracture (open, closed, monolateral or bilateral) requiring surgical intervention and be eligible for fixation by intramedullary nailing. Patients with delayed treatment (initial treatment by external fixation due to swelling / high energy trauma followed by definitive treatment by intramedullary nail) can also be included.
* Patient has been or is scheduled to be treated with the ZNN Bactiguard System Retrograde Femoral Nail.
* Patient must be able and willing to complete the protocol required follow-up.
* Patient must have a signed EC approved consent.
* Patients capable of understanding the surgeon's explanations and following his instructions.

Exclusion Criteria:

* Skeletally immature patients
* A medullary canal obliterated by a previous fracture or tumor
* Bone shaft having excessive bow or a deformity
* Lack of bone substance or bone quality, which makes stable seating of the implant impossible
* All concomitant diseases that can impair the operation, functioning or the success of the implant
* Insufficient blood circulation
* Infection
* Patient is unwilling or unable to give consent.
* Patient is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, alcohol/drug addiction, known to be pregnant or breast feeding).
* Patient anticipated to be non-compliant and/or likely to have problems with maintaining follow-up program (e.g. patient with no fixed address, long distance, plans to move during course of study).
* Not expected to survive the duration of the follow-up program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of 18-year-old patients or older with femur fractures implanted with a ZNN Bactiguard Retrograde Femoral Nail according to the approved/cleared indications.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of fracture healing 12 months after fracture fixation | 3, 6, and 12 months after fracture fixation
  Fracture healing is assessed with x-ray imaging and clinical examination.
  Radiographic Union-Scale in Tibial fractures (RUST) score adapted for the femur, A/P and lateral views. Range: 4 - 12. Fracture healing is defined as RUST scores greater than or equal to 6.
  Fix-IT score (clinical examination). Range 0 - 12, higher scores indicate better limb function.

SECONDARY OUTCOMES:
Oxford Knee Score (limb function) | 3, 6, and 12 months after fracture fixation
  Range: 0 - 48, higher scores indicate better function. Patient-reported outcome to evaluate the function of the limb treated with ZNN Bactiguard Femur Retrograde.
EQ-5D-5L score (patient's quality of life) | pre-surgery (retrospectively), 3, 6, and 12 months after fracture fixation
  Range: 0 - 100, higher scores indicate better quality of life. Patient-reported outcome to evaluate quality of life.
Adverse events frequency | 12 months after fracture fixation
  The incidence and frequency of adverse events occurring during the study will be reported.
Rate of fracture-related infections | 12 months after fracture fixation
  Fracture-related infections are diagnosed in accordance with the algorithm described in M McNally,G Govaert, M Dudareva, M Morgenstern, W J Metsemakers, EFORT Open Rev 2020;5:614-619.

CONTACTS AND LOCATIONS:
Locations (4):
- Hospital Universitario Ntra. Sra. de Candelaria, Santa Cruz de Tenerife, Tenerife, Spain
- United Kingdom (3):
  - Leeds General Infirmary, Leeds, LEEDS
  - Manchester Royal Infirmary, Manchester
  - Stepping Hill Hospital, Stockport